CLINICAL TRIAL: NCT05174442
Title: A Registry-based, Multicenter, International, Post Market Follow-up Study to Monitor the Safety, Performance and Usability of Occlutech Accessory Medical Devices:Occlutech Delivery Set (ODS), Occlutech Pistol Pusher (OPP), Occlutech Occlusions-Pusher (OOP), Occlutech Sizing Balloon (OSB) Used During to Implantation Procedures of Cardiac Implant Devices
Brief Title: ACCESS Registry: A Post Market Follow-up Study to Monitor the Safety, Performance and Usability of Occlutech Accessory Medical Devices
Status: Recruiting | Type: Observational
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Occ2021_03
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-07

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The registry is an international, multicenter, non-randomized, non-invasive study to assess the safety, performance and usability of the Occlutech Accessories "Occlutech Delivery Set (ODS), Occlutech Pistol Pusher (OPP), Occlutech Occlusions-Pusher (OOP) and Occlutech Sizing Balloon (OSB)" used for implantation procedures (catheter-based interventions) of cardiac implants via completing surveys (questionnaires) for the accessory medical devices by the investigators.

DETAILED DESCRIPTION:
The registry is an international, multicenter, non-randomized, non-invasive study to assess the safety, performance and usability of the Occlutech Accessories "Occlutech Delivery Set (ODS), Occlutech Pistol Pusher (OPP), Occlutech Occlusions-Pusher (OOP) and Occlutech Sizing Balloon (OSB)" used for implantation procedures (catheter-based interventions) of cardiac implants via completing surveys (questionnaires) for the accessory medical devices by the investigators.

A survey (questionnaire) of each accessory medical device should be completed by investigator in order to assess safety of the accessory by success of implantation procedure, occurrence of adverse events during implantation procedure or as late term effects resulting from implantation procedure, user harm related to the accessory, procedure, reported device deficiencies related to the accessory. The Surveys (questionnaires) also include questions related to performance, usability and compatibility with devices and other accessories. Subjects should be treated according to instructions-for-use of the implants and accessories and according to clinical routine. The devices must have been used exclusively by physicians who are experienced in cardiac catheterization techniques and who are experienced in using the products in the process of interventional operations.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria depend exclusively on the requirements outlined in the applicable Instruction for Use for accessory medical devices and cardiac implant devices.

All subjects who underwent implantation procedure with an Occlutech accessory medical device and cardiac implants can be included

Exclusion Criteria:

* Exclusion Criteria depend exclusively on the requirements outlined in the applicable Instruction for Use and if applicable in the corresponding protocol of the investigation on the Occlutech implant devices.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects who underwent implantation procedure with an Occlutech accessory medical device and cardiac implants can be included. Preconditions depend exclusively on the requirements outlined in the applicable Instruction for Use of the implant and the accessories.
Sampling Method: Probability Sample
Enrollment: 685 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Occurence of safety events | 6 months
  The primary safety endpoint is defined as the rate of incidences of (peri-) procedural adverse events / rate of (serious) adverse device effects ((S)ADEs) during implantation or as late effects of implantation procedure. A serious adverse device effect (SADE) is defined as an event that is clearly caused by the device such as:
  * device dislocation (during the procedures with OPP, OOP,ODS)
  * embolization related with procedure and accessories
  * Late effect of implantation procedure: damage to the vessels and heart caused by the accessories
  * any circumstances that require device removal related with procedure or accessories used during the implantation
  * Signs of thrombosis

SECONDARY OUTCOMES:
Performance, usability: | 6 months
  will be assessed in terms of mechanical performance, procedural data by completing the survey (questionnaire) for each accessory with grading. Compatibility of ODS, OPP, OOP with cardiac implant devices or/and other accessory medical devices.

CONTACTS AND LOCATIONS:
Locations (35):
- Germany (3):
  - Universitätsklinikum Erlangen, Erlangen
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Klinikum der Universität München, München
- Turkey (Türkiye) (32):
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi, Adana, Balcalı
  - İnönü Üniversitesi Tıp Fakültesi Hastanesi, Malatya, Battalgazi
  - İzmir Şehir Hastanesi, Izmir, Bayraklı
  - Aydın Adnan Menderes Üniversitesi Hastanesi, Aydin, Efeler
  - Bezmialem Tıp Fakültesi Hastanesi, Istanbul, Fatih
  - Antalya Akdeniz Üniversitesi Hastanesi, Antalya, Konyaaltı
  - İstanbul Mehmet Akif Ersoy Göğüs Kalp ve Damar Cerrahisi Eğitim ve Araştırma Hastanesi, Istanbul, Küçükçekmece
  - Karaman Eğitim ve Araştırma Hastanesi, Karaman, Merkez
  - Dicle Üniversitesi Tıp Fakültesi Hastanesi, Diyarbakır, Sur
  - Medicana International Ankara Hastanesi, Ankara, Söğütözü
  - Ankara Etlik Şehir Hastanesi, Ankara, Yenimahalle
  - Adana City Training and Research Hospital, Adana
  - Hacettepe Üniversitesi Hastanesi, Ankara
  - Gazi University Medical Faculty Hospital Adult, Ankara
  - Gazi University Medical Faculty Hospital Pediatric, Ankara
  - Antalya Training and Research Hospital (Adult), Antalya
  - Antalya Training and Research Hospital (Pediatric), Antalya
  - SBÜ Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa
  - Pamukkale Üniversitesi Klinik Uygulama ve Araştırma Merkezi Hastanesi, Denizli
  - Dicle Üniversitesi Tıp Fakültesi Sağlık ve Araştırma Hastanesi, Diyarbakır
  - Eskişehir Osmangazi University Adult, Eskişehir
  - Eskişehir Osmangazi University Pediatric, Eskişehir
  - Isparta Süleyman Demirel Üniversitesi Araştırma ve Uygulama Hastanesi, Isparta
  - Istanbul Basaksahir Cam and Sakura City Hospital(Adult), Istanbul
  - Istanbul Basaksehir Cam and Sakura City Hospital (Pediatric), Istanbul
  - Istanbul Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Kocaeli University Hospital, Kocaeli
  - Necmettin Erbakan Üniversitesi Meram Tıp Fakültesi, Konya
  - Mardin Artuklu Üniversitesi Tıp Fakültesi Hastanesi, Mardin
  - Mersin University Faculty of Medicine Hospital, Mersin
  - S.B.Ü Ahi Evren Göğüs Kalp ve Damar Cerrahisi Eğitim ve Araştırma Hastanesi, Trabzon
  - Gaziantep Üniversitesi Şahinbey Araştırma ve Uygulama Hastanesi, Gaziantep, Şehitkamil